CLINICAL TRIAL: NCT00289328
Title: Glucocorticoid-induced Osteopenia in Children
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Other Study IDs: DK60030 (completed)
Record Dates: First submitted 2006-02-08; First posted 2006-02-09 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Crohn's Disease; Nephrotic Syndrome
MeSH Terms: conditions — Crohn Disease; Nephrotic Syndrome

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to characterize the skeletal deficits and risk factors for impaired skeletal development in children requiring glucocorticoid therapy.

We will compare the bone health of children treated with prednisone for nephrotic syndrome (NS with those treated with prednisone for Crohn's Disease (CD). Childhood NS usually responds to prednisone and is not characterized by pathologies that can impact on bone. In contrast, CD is treated with prednisone, but is independently associated with poor growth and maturation, nutritional deficiencies and inflammation. Due to the differences in the diseases, this comparison will allow us to distinguish between the prednisone-related and disease-related effects on bone in the two disease states.

DETAILED DESCRIPTION:
Prednisone, a glucocorticoid medication, is widely used for many pediatric disorders. Studies have shown that this drug decreases bone formation, decreasing bone density and bone thickness in children. Prednisone induced osteopenia, or low bone density, can be worsened by the effects of the underlying disease, such as delayed growth and maturation, malnutrition, and increased bone resorption (removal) by inflammatory compounds. The combined effects of decreased bone formation and increased resorption may be particularly detrimental to the growing skeleton.

Subjects will include 15 newly diagnosed NS patients, 60 patients with pre-existing NS, 90 patients with newly diagnosed CD, 45 patients diagnosed within the last two years and 200 healthy controls of similar age, gender and ethnicity. Participants will visit the Children's Hospital of Philadelphia (CHOP) three times over a 12-month period for assessment of bone mineralization and turnover, fracture history, dietary calcium intake, physical activity, growth, body composition, muscle strength and glucocorticoid exposure.

ELIGIBILITY:
Inclusion Criteria:

* ages 5-21
* clinical and pathological diagnosis of Crohn's Disease within the last 2 years
* clinical diagnosis of nephrotic syndrome and taking corticosteroids within the last year
* normal renal function GFR>75 ml/min/1.73m2
* healthy controls

Exclusion Criteria:

* other major medical conditions affecting growth and/or bone health
* significant cognitive or developmental disorders (if child is unable to cooperate sufficiently)
* nonambulatory

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 550
Dates: Start 2001-11; Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary B Leonard, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States